CLINICAL TRIAL: NCT04961346
Title: Sublay Technique With Retromuscular Mesh Augmentation for Incisional Hernia Repair - A Prospective Randomized Multicentre Trial Comparing "Lightweight" Versus "Heavyweight" Meshes
Brief Title: RCT Comparing Lightweight vs. Heavyweight Meshes in Incisional Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Andreas Kroh, MD, Principal Investigator, RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ultrapo-Studie
Record Dates: First submitted 2021-06-16; First posted 2021-07-14 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrapro® (Experimental): Participants received incisional hernia repair with an Ultrapro mesh in a sublay technique.
  Interventions: Device: Ultrapro® mesh
- Premilene® (Experimental): Participants received incisional hernia repair with a Premilene mesh in a sublay technique.
  Interventions: Device: Premilene® mesh

INTERVENTIONS:
Device: Ultrapro® mesh — large-pore, lightweight polypropylene mesh
  Arms: Ultrapro®
Device: Premilene® mesh — small-pore, heavyweight polypropylene mesh
  Arms: Premilene®

SUMMARY:
In this randomized, controlled, prospective multicentre clinical trial with a parallel group design a large-pore, lightweight polypropylene mesh (Ultrapro®) is compared to a small-pore, heavyweight polypropylene mesh (Premilene®), within a standardized, retromuscular mesh augmentation to identify the superiority of the lightweight mesh. Included patients are examined at five scheduled follow-up visits (5 and 21 days, 4, 12 and 24 months after surgery). The primary outcome criterion is foreign body sensation 12 month after surgery. Further secondary endpoint criteria are the occurrence of haematoma or haematoma requiring surgery at the 5-day visit, seroma, wound infection, and chronic pain within 24 months postoperatively. Quality of life was investigated by the SF-36®.

ELIGIBILITY:
Inclusion Criteria:

* fascial defect after vertical midline laparotomy with a minimum of 4 cm in diameter

Exclusion Criteria:

* hernia of other location
* recurrent hernia
* incarcerated hernia
* emergency surgery
* patients with a malignancy or chemotherapy within the last 3 months
* pregnancy
* participation in other studies
* patients with a wound infection
* missing informed consent

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2007-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
foreign body sensation | 12 month after surgery
  Quality of life measurement based on the occurrence of a foreign body sensation for more than 3 months within 12 month after surgery.

SECONDARY OUTCOMES:
postoperative seroma | 24 month
  Fluid collection in the wound area
wound infection | 24 month
  Clinical identification of superficial and deep wound infections.
haematoma | 5 days
  hematoma in the wound area
hematoma requiring surgery | 5 days
  hematoma in the wound area requiring surgery
chronic pain | 24 month
  Chronic pain is defined as pain sensations that persist for more than 3 months after surgery. A Visual Analog Scale (VAS) with a range of 0-10 is used as a tool to measure pain.
hernia recurrence | 24 month
  hernia recurrence is defined as a new abdominal wall defect in the area of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ralf D Hilgers, Professor, Principal Investigator — Institute for Medical Statistics, RWTH Aachen University Hospital, Aachen, Germany
Locations (1):
- Department of Surgery, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kroh A, Zufacher M, Eickhoff R, Heise D, Helmedag M, Ulmer F, Neumann UP, Conze J, Hilgers RD, Binnebosel M. No difference in outcomes between large- and small-pore meshes in a prospective, randomized, multicenter trial investigating open retromuscular meshplasty for incisional hernia repair. Langenbecks Arch Surg. 2023 Jan 13;408(1):22. doi: 10.1007/s00423-022-02751-x. PMID 36635466